CLINICAL TRIAL: NCT02050386
Title: The Role of Brain Arousal Systems in Cognitive and Physical Decline in Normal Aging
Brief Title: The Brain Alerting Mechanism Study
Status: Withdrawn | Type: Observational
Why Stopped: Resources were refocused into another project preventing this project from starting
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201300392
Record Dates: First submitted 2014-01-23; First posted 2014-01-30 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Healthy Volunteers
Keywords: Brain arousal systems; Aging; MRI; fMRI; Cognition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cold pressor stimulation: Immersion of the foot in 0-2 degrees C water for 50 seconds.
  Interventions: Other: Cold pressor stimulation
- Sham Stimulation: Immersion of the foot in room temperature water for 50 seconds.
  Interventions: Other: Sham Stimulation

INTERVENTIONS:
Other: Cold pressor stimulation — Immersion of the foot in 0-2 degrees C water for 50 seconds
  Groups: Cold pressor stimulation
Other: Sham Stimulation — Immersion of the foot in room temperature water for 50 seconds
  Groups: Sham Stimulation

SUMMARY:
This is a study designed to look at how arousal levels in the brain change with age and how these changes influence thinking, vision, hearing and physical function in people of advanced age.

DETAILED DESCRIPTION:
There are two parts involved in this study:

Part #1- Paperwork, Computer-based cognitive tests, Physical function test, EEG recording

* Potential participants will be pre-screened at the time of their initial phone call to be sure they fit the guidelines for this research study.
* Participants will be given this Informed Consent document. This Informed Consent will be reviewed in a private location; participants will be given as much time as participants need to consider enrolling in the study. Participants may want to discuss the information with friends or family. Participants may ask questions at any time during the study visit.
* If participants choose to sign this form, and agree to participate, participants will be further screened for inclusion/exclusion factors related to the MRI scanning. All women under the age of 62 will be given a pregnancy test, based on a urine sample.
* Investigators will review a detailed Medical History form with participants, asking questions about participants and participants family's medical history.
* Investigators will ask participants to complete a brief physical activity questionnaire asking questions about participants daily level of physical activity.
* Participants will be asked to complete several computer tasks meant to measure participants cognitive abilities (like memory and attention), which takes about 30 minutes.
* Participants will also be asked to complete a short physical performance battery (SPPB), that looks at participants ability to sit and stand, walk a short distance, and balance, which takes about 30 minutes.
* Participants will also be asked to participate in an EEG recording session. An EEG cap, selected for participants head size, will be placed on participants head. The cap contains small electrodes that record participants brains electrical activity. During this part of the study, participants will sit in a comfortable chair while watching pictures on a computer screen, listening to sounds through headphones, or resting. This will take about 1 hour.
* Participants will also be asked to undergo a cold pressor test (CPT) and/or sham stimulation. CPT involves immersing either participants hand or foot in cold water for about one minute. Sham stimulation involved immersing either the hand or foot in room temperature water for about one minute.
* Finally, participants will be transported by someone involved with this study (by passenger van or golf cart) to the McKnight Brain Institute MRI Center. Or, if participants prefer, the next portion of the visit can be scheduled for another day.

Part #2- MRI Scan

The following procedures will take place at the Advanced Magnetic Resonance Imaging Center at the McKnight Brain Institute- for the MRI brain scan, and can be done on the same day as Part #1, or on a different day for participants scheduling convenience.

Magnetic resonance imaging (MRI) is a procedure that allows doctors to look inside the body by using a scanner that sends out a strong magnetic field and radio waves. This procedure is used routinely for medical care and is very safe for most people, but participants will be monitored during the entire MRI scan in case any problems occur. The risks of MRI are:

* The MRI scanner contains a very strong magnet. Therefore, participants may not be able to have the MRI if participants have any type of metal implanted in participants body, for example, any pacing device (such as a heart pacer), any metal in participants eyes, or certain types of heart valves or brain aneurysm clips. Someone will ask participants questions about this before participants have the MRI.
* There is not much room inside the MRI scanner. Participants may be uncomfortable if participants do not like to be in close spaces ("claustrophobia"). During the procedure, participants will be able to talk with the MRI staff through a speaker system, and, in the event of an emergency, participants can tell them to stop the scan.
* The MRI scanner produces a loud hammering noise, which has produced hearing loss in a very small number of patients. Participants will be given earplugs to reduce this risk.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 95

Exclusion Criteria:

* History of pre-existing neurological disorders,
* Psychiatric brain disorders,
* Diagnosis with a neurodegenerative brain disease,
* Uncontrolled blood pressure (>200/110),
* History of severe hypertension,
* History of angina
* People who have metal implants and can not have an MRI scan,
* People who are claustrophobic,
* Females of child-bearing age and have a positive test for pregnancy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults 18 and older.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Cognitive Function | Baseline
  The Cognition Domain measures several aspects of cognitive functioning for ages 3-85, including language, episodic memory, executive function, working memory and processing speed.
  To interpret individual performance, one can evaluate all three types of scale scores. A participant's age-adjusted scale score at or near 100 indicates vocabulary ability that is average for the age level. Scores around 115 suggest above-average vocabulary ability, while scores around 130 suggest superior ability.
MRI: BOLD Response | Baseline
  Functional MRI
Cognitive Function | up to 30 days
  The Cognition Domain measures several aspects of cognitive functioning for ages 3-85, including language, episodic memory, executive function, working memory and processing speed.
  To interpret individual performance, one can evaluate all three types of scale scores. A participant's age-adjusted scale score at or near 100 indicates vocabulary ability that is average for the age level. Scores around 115 suggest above-average vocabulary ability, while scores around 130 suggest superior ability.
MRI: BOLD Response | up to 30 days
  Functional MRI

SECONDARY OUTCOMES:
Physiological Response: Mean Heart Rate | Baseline
  Heart Rate
Cognitive Functions: N-Back Task Test | Baseline
  N-Back Score is as follows: the mean is 100 and the standard deviation (SD) is 15.
Cognitive Functions: Attention Tasks Test | Baseline
  Attention tests score is measured using a of mean 100 and the standard deviation (SD) is 15.
Cognitive Functions: Memory Task Test | Baseline
  The memory tests scoring for ease of understanding, corresponds to an Age-Adjusted Scale Score of 115 - exactly 1 SD above the mean of 100.
Physical Function: Short Physical Performance Battery | Baseline
  Short battery of tests that include walking and standing. The score includes the distance to range from 400m to 700m. A lower score indicates worse function.

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Woods, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States